CLINICAL TRIAL: NCT06114043
Title: Randomised Controlled Trial; Is Operative Treatment of Mild to Moderate Hallux Valgus Deformity Superior to Conservative Treatment?
Brief Title: Operative Versus Non-operative Treatment for Mild to Moderate Hallux Valgus Deformity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Marius Molund, MD, phd, head of foot & ankle department Ostfold hospital trust, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 575297
Record Dates: First submitted 2023-03-20; First posted 2023-11-02 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hallux Valgus Deformity
MeSH Terms: interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial investigating patients with painful mild to moderate hallux valgus deformity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operation (Other): 60 participants will be operated for mild to moderate hallux valgus deformity
  Interventions: Other: Operation for mild to moderate hallux valgus
- Conservative (Other): 60 participants will be treated conservatively with a wide shoe
  Interventions: Other: Conservative treatment with orthopedic aid/wide shoe for participants with mild to moderate hallux valgus

INTERVENTIONS:
Other: Conservative treatment with orthopedic aid/wide shoe for participants with mild to moderate hallux valgus — 60 participants will receive conservative treatment with orthopedic aid/wide shoe. Participants will be followed for 2 years.
  Arms: Conservative
Other: Operation for mild to moderate hallux valgus — 60 participants will receive the traditional operative treatment for the deformity. Participants will be followed for 2 years.
  Arms: Operation

SUMMARY:
The goal of this randomized controlled trial is to investigate operative treatment versus conservative treatment in participants suffering from mild to moderate hallux valgus deformity. The main question it aims to answer are; Is surgery superior to conservative treatment?

The participants will be randomized in to two groups, operative and conservative group.

Investigators will compare the groups measuring the clinical results using the patient-reported outcome measure (PROM) Manchester-Oxford Foot Questionnaire (MOxFQ), Visual analog scale (VAS), likert scale 0-5. Participants will be observed for a period og two years.

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) investigating the patient reported outcome after operative or conservative treatment in mild to moderate hallux valgus deformity. In this RCT study participants will be divided into operative group, non-operative group where the treatment will be orthopedic aids/wide shoes. The participants will be evaluated 6 months, 1 year and 2 years after starting the treatment. The clinical results will be evaluated using patient reported outcome measures (PROMs).

Primary aim: Investigating the clinical result by PROM (Manchester Oxford Foot Questionnaire)

Secondary aim: Investigating the radiological results according to newer and traditional parameters. Operative group -correction achieved, residual rate. Conservative group -progression of deformity.

Statistical power calculations have been made within the research group. Calculations are based on the main outcome MOxFQ, with the power of 80 and confidence interval 95%. The investigators concluded that a sample size of 49 participants will be needed to perform a regression analysis. To account for loss to follow-up (estimated 20%),120 participants (60 per group) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Painful Hallux Valgus deformity
* Hallux Valgus Angle <35 degrees
* Intermetatarsal angle <15 degrees
* 18-80 years

Exclusion Criteria:

* Advanced osteoarthritis in first metatarsophalangeal joint
* Rheumatic diseases
* Pregnancy
* Drug abuse
* Severe psychological disorder
* Lack of compliance
* Language barrier

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Clinical results MOxFQ | 2 years
  Manchester oxford foot questionnaire (MOxFQ) (Raw scores can be converted to a 0-100 metric where 100=most severe)

SECONDARY OUTCOMES:
Clinical result VAS | 2 years
  Visual analogue scale (VAS) 0-10 (0=best to 10=worst)
Clinical result SF-36 | 2 years
  Short Form Health Survey (SF-36) (0=worst to 100=best)
Clinical result Likert scale | 2 years
  Likert scale 0-5 (0=worst to 5=best)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: No